CLINICAL TRIAL: NCT04635644
Title: Ultrasound Guided Erector Spinae Block Versus Intrathecal Morphine for Postoperative Analgesia in Major Hepatopancreaticobiliary Surgery
Brief Title: Ultrasound Guided ESP Block Versus Intrathecal Morphine for Postoperative Analgesia in Major HPB Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Magdy Mohammed Mahdy Sayed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ABC-4-DE
Record Dates: First submitted 2020-11-14; First posted 2020-11-19 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): Patients will receive Erector spinae plane block.
  Interventions: Procedure: Erector Spinae Plane Block
- Intrathecal morphine ITM (Active Comparator): Patients will receive Intrathecal morphine.
  Interventions: Procedure: Intrathecal morphine

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Patients will be turned into the prone position. A high-frequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation 2.5-3 cm lateral to the T8 spinous process. The erector spinae muscles will be identified superficial to the tip of the T8 transverse process. After local infiltration of the needle insertion site with 2-3 ml of 2% lidocaine, a 21G 10 cm needle will be inserted using an in-plane approach in a cranial to caudal direction to contact the T8 transverse process. The location of the needle tip will be confirmed by hydrodissection with 2 mL of lidocaine 2% and visualizing linear fluid spread lifting the erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging. A volume of 20 mL of 0.25% Bupivacaine is injected will be injected at this point. The same procedure will be repeated for the opposite side.
  Other Names: ESP block
  Arms: Erector Spinae Plane Block
Procedure: Intrathecal morphine — Patients will be placed on their right side. An intrathecal injection of morphine 200 μg (0.2 mL of morphine sulfate 1 mg/mL) diluted in 1.8 mL normal saline will be administered at the L3-L4 or L4-L5 level with a 25 G Whitacre spinal needle.
  Other Names: ITM
  Arms: Intrathecal morphine ITM

SUMMARY:
To compare the efficacy of USG-guided bilateral Erector spinae plane block (ESPB) with intrathecal morphine (ITM) for postoperative analgesia after major hepatopancreaticobiliary surgery (HPB)

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years with a body mass index (BMI) of 18-35 kg/m2,
* patients with the American Society of Anesthesiologists (ASA) physical status I - II,
* Patients scheduled for elective major hepatopancreaticobiliary surgery for benign or malignant disease; major surgery is defined as an operation of anticipated duration of more than one hour.

Exclusion Criteria:

* Patient's refusal
* Allergy or contraindications to the study drugs,
* Infection at the site of injection,
* Coagulopathy,
* Psychiatric disorders
* Severely co-morbid patients,
* Chronic pain syndromes,
* Prolonged opioid medication,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Cumulative opioid consumption | 24 hours postoperatively
  Nalbuphine consumption in mg equivalent to morphine dose

SECONDARY OUTCOMES:
Nalbuphine consumption in mg | at 8, 48, and 72 hours postoperatively.
  equivalent to morphine dose
Analgesic drug consumption other than nalbuphine | at 8, 24, 48, and 72 hours postoperatively.
  consumption in mg
Numerical Rating Scale (NRS) at rest and when coughing | at 1, 2, 4, 8, 12, 24, 48 and 72 hours postoperatively
  NRS is an 11-point (0=no pain and 10=worst pain)
Heart Rate | Intraoperatively
  Heart Rate in beats /min
Mean Arterial Pressure | Intraoperatively
  Mean Arterial Pressure in mmHg
Incidence of Postoperative nausea & vomiting (PONV) | 24 hours postoperatively
  Number of patients developing PONV

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt